CLINICAL TRIAL: NCT02305316
Title: Single-dose Pharmacokinetics and Relative Bioavailability of Two Different Formulations of Opicapone in Healthy Volunteers
Brief Title: Single-dose Pharmacokinetics and Relative Bioavailability of Two Different Formulations of Opicapone
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bial - Portela C S.A. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: BIA-91067-120
Record Dates: First submitted 2014-11-28; First posted 2014-12-02 (Estimated); Results first posted 2015-08-21 (Estimated); Last update posted 2015-08-21 (Estimated); Status verified 2015-07

CONDITIONS: Parkinson Disease
MeSH Terms: conditions — Parkinson Disease | interventions — opicapone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- BIA 9-1067 non-micronized - micronized (Experimental): Each subject was orally administered with 50 mg OPC non-micronized followed by a washout period of 14 days. After washout period each subject was orally administered with 50 mg OPC micronized
  Interventions: Drug: BIA 9-1067 non-micronized; Drug: BIA 9-1067 micronized
- BIA 9-1067 micronized - non-micronized (Experimental): Each subject was orally administered 50 mg OPC micronized followed by a washout period of 14 days. After washout period each subject was orally administered with 50 mg OPC non-micronized
  Interventions: Drug: BIA 9-1067 non-micronized; Drug: BIA 9-1067 micronized

INTERVENTIONS:
Drug: BIA 9-1067 non-micronized
  Other Names: OPC, Opicapone
Drug: BIA 9-1067 micronized
  Other Names: OPC, Opicapone

SUMMARY:
Single-centre, open-label, randomised, two-way crossover study in 28 healthy volunteers. The study consisted of two consecutive single-dose treatment periods separated by a washout period of 14 days or more.

DETAILED DESCRIPTION:
Single-centre, open-label, randomised, two-way crossover study in 28 healthy volunteers. The study consisted of two consecutive single-dose treatment periods separated by a washout period of 14 days or more. A total of twenty-eight (28) healthy volunteers received a single dose of 50 mg OPC, orally.

ELIGIBILITY:
Inclusion Criteria:

* A signed and dated informed consent form (ICF) before any study-specific screening procedure was performed,
* Male or female subjects aged 18 to 45 years, inclusive,
* Body mass index (BMI) between 19 and 30 kg/m2,
* Healthy as determined by pre-study medical history, physical examination, vital signs, complete neurological examination and 12-lead electrocardiogram (ECG),
* Negative tests for hepatitis B surface antigen (HBsAg), anti-hepatitis C virus (HCV) antibodies and anti-human immunodeficiency virus (HIV) antibodies at screening,
* Clinical laboratory test results clinically acceptable at screening and on D-1 of each treatment period,
* Negative screen for alcohol and drugs of abuse at screening and on D-1 of each treatment period,
* Non-smokers or ex-smokers for at least 3 months,
* Volunteer able to participate, and willing to give written informed consent and comply with the study restrictions,

If female:

* Was not of childbearing potential by reason of surgery or, if of childbearing potential, uses an effective non-hormonal method of contraception (intrauterine device or intrauterine system; condom or occlusive cap [diaphragm or cervical or vault caps] with spermicidal foam or gel or film or cream or suppository; true abstinence; or vasectomized male partner, provided that he was the sole partner of that subject) for the entire duration of the study,
* Negative serum pregnancy test at screening and a negative urine pregnancy test on D-1 of each treatment period.

Exclusion Criteria:

* Any clinically relevant history or presence of respiratory, gastrointestinal, renal, hepatic, haematological, lymphatic, neurological, cardiovascular, psychiatric, musculoskeletal, genitourinary, immunological, dermatological, endocrine, connective tissue diseases or disorders, or had a clinically relevant surgical history,
* Any clinically relevant abnormality in the coagulation tests,
* Any clinically relevant abnormality in the liver function tests,
* History of relevant atopy or drug hypersensitivity,
* History of alcoholism and/or drug abuse,
* Current consumption of more than 14 units of alcohol per week [1 unit of alcohol = 280 mL beer (3-4°) = 100 mL wine (10-12°) = 30 mL spirits (40°)],
* Any significant infection or known inflammatory process on screening or admission to each treatment period,
* Any acute gastrointestinal symptoms (e.g., nausea, vomiting, diarrhoea, heartburn) at the time of screening or admission to each treatment period,
* Use of medicines within 2 weeks of admission to first period that could affect the subject's safety or other study assessments, in the investigator's opinion,
* Previously received opicapone,
* Involvement in other clinical trials of any type within 90 days prior to screening,
* Participation in more than 2 clinical trials within the 12 months prior to screening,
* Blood donation or received any blood transfusion or any blood products within the 3 months prior to screening,
* Vegetarian, vegan or had medical dietary restrictions,
* Subject not able to communicate reliably with the investigator,
* Subjects who were unlikely to co-operate with the requirements of the study,
* Subjects who were unwilling or unable to give written informed consent,

If female:

* Pregnant or breast-feeding,
* If of childbearing potential, a positive serum pregnancy test,
* Volunteer who did not use an accepted effective contraceptive method or used oral contraceptives,

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 28 (Actual)
Dates: Start 2014-02; Primary Completion 2014-03 (Actual); Study Completion 2014-03 (Actual)

RESULTS

PARTICIPANT FLOW:
Groups:
- BIA 9-1067 Non-micronized - Micronized: Each subject was orally administered with 50 mg OPC non-micronized followed by a washout period of 14 days. After washout period each subject was orally administered with 50 mg OPC micronized
  BIA 9-1067 non-micronized
  BIA 9-1067 micronized
- BIA 9-1067 Micronized - Non-micronized: Each subject was orally administered 50 mg OPC micronized followed by a washout period of 14 days. After washout period each subject was orally administered with 50 mg OPC non-micronized
  BIA 9-1067 non-micronized
  BIA 9-1067 micronized
Period: Overall Study
Arm/Group | BIA 9-1067 Non-micronized - Micronized | BIA 9-1067 Micronized - Non-micronized
Started | 14 | 14
Completed | 14 | 14
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | BIA 9-1067 Non-micronized - Micronized | BIA 9-1067 Micronized - Non-micronized | Total
Number analyzed (Participants) | 14 | 14 | 28
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 14 | 14 | 28
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 7 | 14
  Male | 7 | 7 | 14

OUTCOME MEASURES:

1. Primary Outcome: Cmax - Maximum Observed Plasma Concentration
Description: Maximum observed plasma concentration of BIA 9-1067
Time Frame: before OPC dosing, and 0.5, 1, 2, 3, 4, 6, 8, 12, 16, 24, 36 and 48 hours post-OPC dose.
Measure: Mean (Standard Deviation); unit: ng/mL
Groups:
- BIA 9-1067 Non-micronized: BIA 9-1067 non-micronized.
- BIA 9-1067 Micronized: BIA 9-1067 micronized.
Arm/Group | BIA 9-1067 Non-micronized | BIA 9-1067 Micronized
Number analyzed (Participants) | 28 | 28
ng/mL | 327.8 (129.6) | 750.1 (184.1)

2. Secondary Outcome: AUC0-t - Area Under the Plasma Concentration-time Curve From Time 0 to the Time of Last Quantifiable Concentration
Description: AUC0-t - Area under the plasma concentration-time curve from time 0 to the time of last quantifiable concentration of BIA 9-1067
Time Frame: before OPC dosing, and 0.5, 1, 2, 3, 4, 6, 8, 12, 16, 24, 36 and 48 hours post-OPC dose.
Measure: Mean (Standard Deviation); unit: ng.h/mL
Arm/Group | BIA 9-1067 Non-micronized | BIA 9-1067 Micronized
Number analyzed (Participants) | 28 | 28
ng.h/mL | 1152.8 (537.5) | 2296.5 (778.2)

3. Secondary Outcome: Tmax - Time of Occurrence of Cmax of BIA 9-1067
Description: tmax - time of occurrence of maximum observed plasma concentration of BIA 9-1067
Time Frame: before OPC dosing, and 0.5, 1, 2, 3, 4, 6, 8, 12, 16, 24, 36 and 48 hours post-OPC dose.
Measure: Mean (Full Range); unit: hours
Arm/Group | BIA 9-1067 Non-micronized | BIA 9-1067 Micronized
Number analyzed (Participants) | 28 | 28
hours | 2.50 [1.00 to 6.00] | 2.00 [1.00 to 4.00]

4. Secondary Outcome: AUC0-inf - Area Under the Plasma Concentration-time Curve From Time 0 to the Infinity
Description: AUC0-inf - Area under the plasma concentration-time curve from time 0 to the infinity.
Time Frame: before OPC dosing, and 0.5, 1, 2, 3, 4, 6, 8, 12, 16, 24, 36 and 48 hours post-OPC dose.
Measure: Mean (Standard Deviation); unit: ng.h/mL
Arm/Group | BIA 9-1067 Non-micronized | BIA 9-1067 Micronized
Number analyzed (Participants) | 28 | 28
ng.h/mL | 1327.0 (562.0) | 2324.1 (781.8)

ADVERSE EVENTS:
Arm/Group | BIA 9-1067 Non-micronized | BIA 9-1067 Micronized
Serious Adverse Events (participants affected / at risk) | 0/28 | 0/28
Other Adverse Events (participants affected / at risk) | 2/28 | 1/28
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | BIA 9-1067 Non-micronized (N=28) | BIA 9-1067 Micronized (N=28)
Headache (Nervous system disorders) | 2 | 0
Stiff neck (Musculoskeletal and connective tissue disorders) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other